CLINICAL TRIAL: NCT06282445
Title: Efficacy and Safety of Chemotherapy With XELOX (Oxaliplatin + Capecitabine) and Bevacizumab in Combination With Adebrelimab in First-line Treatment of Microsatellite Stable (MSS) Initially Unresectable Metastatic Colorectal Cancer: a Prospective, Multicenter, Single-arm Study
Brief Title: Efficacy and Safety of Chemotherapy With XELOX (Oxaliplatin + Capecitabine) and Bevacizumab in Combination With Adebrelimab in First-line Treatment of Microsatellite Stable (MSS) Initially Unresectable Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY-2024-020
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Colorectal Cancer Metastatic
MeSH Terms: interventions — Oxaliplatin; Capecitabine; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chemotherapy With XELOX (Oxaliplatin + Capecitabine) and Bevacizumab in Combination With Adebrelimab (Experimental): The enrolled patients with microsatellite stable (MSS) initially unresectable metastatic colorectal cancer will receive a chemotherapy with XELOX and Bevacizumab in combination with Adebrelimab in first-line treatment.
  XELOX: Oxaliplatin 130 mg/m2, day 1, q3w; Capecitabine 1000 mg/m2, bid, d1-d14, q3w; Bevacizumab: 7.5mg/kg, intravenous infusion, day 1. q3w. Adebrelimab: intravenously guttae, 1200mg, day 1, q3w. 4 cycles.
  Imaging assessment of tumor remission was performed every 8 weeks. Patients who received 4-6 months of treatment and achieved disease control entered the maintenance treatment stage, receiving maintenance treatment:
  Bevacizumab: 7.5mg/kg, intravenous infusion, d1, Q3W; Capecitabine: 1250mg/ m2, orally, bid, Q3W; Adebrelimab: 1200mg, intravenous infusion, day 1, Q3W.
  Interventions: Drug: Adebrelimab; Drug: Oxaliplatin; Drug: Capecitabine; Drug: Bevacizumab

INTERVENTIONS:
Drug: Adebrelimab — This product is administered by intravenously guttae. The recommended dose of subcutaneous injection is 1200mg, administered every 3 Weeks (Q3W).
  Other Names: SHR-1316
Drug: Oxaliplatin — 130 mg/m2, ivgtt, d1, Q3W
Drug: Capecitabine — 1000mg/m2, po, bid, d1-14, Q3W Maintenance therapy: 1250mg/m2, po, bid, d1-14, Q3W
Drug: Bevacizumab — 7.5mg/kg，ivgtt, d1, Q3W

SUMMARY:
To evaluate the efficacy and safety of Chemotherapy With XELOX (Oxaliplatin + Capecitabine) and Bevacizumab in Combination With Adebrelimab in First-line Treatment of Microsatellite Stable (MSS) Initially Unresectable Metastatic Colorectal Cancer.

DETAILED DESCRIPTION:
At present, the survival benefit of MSS mCRC patients is limited, and the general survival time is only about 3-4 months. Up to now, the standard treatment plan is FOLFOX combined with bevacizumab. AtezoTRIBE study shows that compared with FOLFOXIRI+ bevacizumab, the standard treatment plan is better than the standard treatment plan. The combination of PD-L1 monomone attillizumab extended mPFS from 11.4 months to 12.9 months, showing certain efficacy, and the combination of Attillizumab did not increase adverse reactions. Based on the above, this study aims to explore the efficacy and safety of chemotherapy with XELOX (oxaliplatin + capecitabine) regimen and bevacizumab combined with adbelizumab in first-line treatment of microsatellite stable (MSS) type of initial unresectable metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1.The patients voluntarily participated in the study, signed the informed consent, and had good compliance.
* 2. Age 18-75 years (including 18 and 75) .
* 3. Metastatic colorectal cancer confirmed histologically and/or cytologically and initially unresectable.
* 4.MSS or pMMR.
* 5.Patients must have at least one measurable lesion (RECIST 1.1).
* 6.ECOG physical condition 0-1 score.
* 7.Expected survival ≥12 weeks.
* 8.Blood examination (no blood transfusion within 14 days, no correction of granulocyte colony stimulating factor or other hematopoietic stimulating factor within 7 days before laboratory examination).

  1. neutrophil absolute value ≥1.5×109/L, platelets ≥100×109/L, hemoglobin concentration ≥9g/dL)
  2. Liver function test (bilirubin ≤1.5×ULN; Aspartate aminotransferase and glutamic acid aminotransferase ≤2.5×ULN, AST and ALT≤5×ULN in the case of liver metastasis);
  3. Renal function (serum creatinine ≤1.5×ULN, or creatinine clearance (CCr)≥60ml/min);
  4. Coagulation, International standardized ratio (INR) ≤1.5×ULN, prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤1.5×ULN;
  5. Thyroid function, thyroid stimulating hormone (TSH) ≤ the upper limit of normal (ULN); If there is any abnormality, FT3 and FT4 levels should be examined. If FT3 and FT4 levels are normal, they can be selected.
* 9.Reproductive-age women must have a negative serum pregnancy test within 14 days before treatment and be willing to use a medically acceptable effective contraceptive method (e.g., an intrauterine device, oral contraceptives, or condoms) during the study and for 3 months after the last study dose; for male subjects who are married to a reproductive-age woman, surgical sterilization is required or effective contraception is recommended during the study and for 3 months after the last study dose.

Exclusion Criteria:

* 1.Received the following treatments within 4 weeks prior to treatment: radiotherapy for tumors, surgery, chemotherapy, immunotherapy or molecular targeted therapy, or other investigational medications.
* 2.Active autoimmune disease requiring systemic therapy (i.e., disease-modifying drugs, corticosteroids, or immunosuppressants) has been used within the past 2 years. Replacement therapies (such as thyroxine, insulin, or physiologic corticosteroid replacement for adrenal or pituitary insufficiency) are not considered systemic therapy.
* 3.Diagnosed with an immune deficiency within 7 days prior to the first treatment or received systemic steroid therapy or any other form of immunosuppressive therapy. The use of physiological doses of corticosteroids may be approved after consultation with the sponsor.
* 4.Previously received anti-vascular small-molecule targeted drug therapy, such as fuquintinib.
* 5.Previous treatment with irinotecan based chemotherapy regimens.
* 6.Symptomatic brain or meningeal metastasis.
* 7.RAS wild-type left half colon cancer.
* 8.Metastatic colorectal cancer with MSI-H or dMMR.
* 9.Severe infection (such as intravenously administered antibiotics, antifungals, or antivirals) within 4 weeks of treatment, or unexplained fever > 38.5 ° C during screening/first administration.
* 10.Have high blood pressure that is not well controlled with antihypertensive medications (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg).
* 11.There were obvious clinical bleeding symptoms or obvious bleeding tendency within 3 months before treatment (bleeding > 30 mL within 3 months, hematemesis, black stool, blood in the stool), hemoptysis (> 5 mL of fresh blood within 4 weeks), etc. Or treatment of venous/venous thrombosis events within the preceding 6 months, such as cerebrovascular accidents (including transient ischemic episodes, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism; Long-term anticoagulant therapy with warfarin or heparin, or long-term antiplatelet therapy (aspirin ≥300 mg/day or clopidogrel ≥75 mg/day) is required.
* 12.During screening, it was found that the tumor invaded large vascular structures, such as pulmonary artery, superior vena cava or inferior vena cava, etc., and the researchers judged that there was a risk of major bleeding.
* 13.Active heart disease, including myocardial infarction, severe/unstable angina, occurred 6 months before treatment. Left ventricular ejection fraction <50% by echocardiography showed poor arrhythmia control.
* 14.Patients have had other malignancies (except cured basal cell carcinoma of the skin and cervical carcinoma in situ) within the previous 5 years or at the same time.
* 15.Is known to be allergic to the investigational drug or any of its excipients.
* 16.Active or uncontrolled severe infection.

  1. Known human immunodeficiency virus (HIV) infection.
  2. Known history of clinically significant liver disease, including viral hepatitis [active HBV infection, i.e., positive HBV DNA (>1×104 copies /mL or >2000IU/ml) must be excluded for known hepatitis B virus (HBV) carriers.
  3. Known hepatitis C virus infection (HCV) and HCV RNA positive (>1×103 copies /mL), or other hepatitis, cirrhosis]

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Up to 2 years
  Progression-free survival (PFS) denotes the chances of staying free of disease progression for a group of individuals suffering from a cancer after a particular treatment.

SECONDARY OUTCOMES:
Organ retention rate | Up to 2 years
  The proportion of patients who achieved pre-specified tumor volume reduction and maintained the minimum time limit was the sum of complete and partial responses.
Overall survival | Up to 2 years
  The proportion of participants who remain survival at 2 years
Disease Control Rate | Up to 2 years
  The percentage of patients with advanced cancer whose therapeutic intervention has led to a complete response, partial response, or stable disease.
Surgical conversion rate | Up to 2 years
  The rate of conversion to surgery.
TRAEs | Up to 2 years
  Number of participants with treatment-related adverse events as assessed by NCI-CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Dezhi Li, MD&PhD, Principal Investigator — China, The Fourth Affiliated Hospital Zhejiang University School of Medicine
Locations (1):
- The Fourth Affiliated Hospital Zhejiang University School of Medicine, Jinhua, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No